CLINICAL TRIAL: NCT01607983
Title: The Effect of Selective Pulmonary Vasodilation on Ventricular Afterload and Ventricular-arterial Coupling in Patients With Fontan Physiology and Validation of Echocardiographic Measures of Systolic and Diastolic Function.
Brief Title: Effects of Pulmonary Vasodilation Upon VA Coupling in Fontan Patients
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Poor accrual
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-06070
Record Dates: First submitted 2012-05-24; First posted 2012-05-30 (Estimated); Last update posted 2018-05-04 (Actual); Status verified 2018-05

CONDITIONS: Congenital Heart Disease; Fontan
Keywords: nitric oxide; ventricular-arterial coupling; congenital heart disease
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- inhaled nitric oxide (Experimental)
  Interventions: Drug: inhaled nitric oxide

INTERVENTIONS:
Drug: inhaled nitric oxide — 20 parts per million (ppm) of inhaled nitric oxide

SUMMARY:
The study involves documenting the effects of inhaled nitric oxide upon ventricular-arterial coupling in patients with congenital heart disease and passive pulmonary blood flow. Consenting patients undergoing a clinically-indicated cardiac catheterization will be given inhaled nitric oxide for 10 minutes while intraventricular pressure-volume analysis will be make via conduction catheters.

DETAILED DESCRIPTION:
Patients with complex congenital heart disease and single ventricle physiology typically undergo a staged surgical palliation to a situation where the single ventricle is recruited as the systemic pumping chamber and some (following a Glenn surgery) or all (following a Fontan surgery) systemic venous return flows passively to the lungs. While this physiology eliminates ventricular volume loading and normalizes systemic arterial oxygen saturations, there remain a number of physiologic burdens that limit functional capacity and life expectancy. Evidence suggests that this surgical imposition of the systemic and pulmonary vascular beds in series results in ventricular loading conditions that adversely affect ventricular function. At present, there exist limited means by which to mitigate these burdens, however, new therapies directed at reducing total pulmonary resistance may favorably affect patients with this physiology by reducing systemic venous pressures and improving both ventricular preload and afterload. One such therapy is inhaled nitric oxide (iNO), which is a selective pulmonary vasodilator that has been shown to reduce total pulmonary resistance and improve systemic venous pressures in this patient population. However limited data exist regarding the affects of pulmonary vasodilators like iNO on ventricular loading and ventricular-arterial coupling. This study proposes to assess the effects of pulmonary vasodilator therapy upon ventricular loading and ventricular-arterial coupling in single ventricle patients with passive pulmonary blood flow presenting for elective cardiac catheterization. The study components include obtaining routine (they would be obtained as a part of the clinically-indicated catheterization) hemodynamic measurements with hi-fidelity catheters rather than standard fluid-filled catheters, as well as simultaneous additional measurements with the same catheters at rest and during administration of iNO.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive patients with single ventricle hearts having passive pulmonary blood flow presenting to the cardiac catheterization laboratory for clinically indicated cardiac catheterization.

Exclusion Criteria:

* Patients with coarctation of the aorta or known bilateral femoral arterial obstruction
* Patients with known severe systemic venous/Fontan obstruction
* Patients already receiving sildenafil or other vasodilator therapy

Ages: 4 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2012-06; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Effective arterial elastance (Ea) | Acute, approximately 10-15 minutes
  Patients will undergo hemodynamic evaluation while receiving inhaled nitric oxide. After the measurements are made the nitric oxide will be discontinued. The primary outcome is the change in effective arterial elastance, a value obtained from ventricular pressure-volume assessment, before and while receiving nitric oxide.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffery Meadows, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Senzaki H, Masutani S, Kobayashi J, Kobayashi T, Sasaki N, Asano H, Kyo S, Yokote Y, Ishizawa A. Ventricular afterload and ventricular work in fontan circulation: comparison with normal two-ventricle circulation and single-ventricle circulation with blalock-taussig shunts. Circulation. 2002 Jun 18;105(24):2885-92. doi: 10.1161/01.cir.0000018621.96210.72. PMID 12070118 (Retraction: PMID 22689940 Circulation. 2012 Jun 12;125(23):e1020)
- [Background] Szabo G, Buhmann V, Graf A, Melnitschuk S, Bahrle S, Vahl CF, Hagl S. Ventricular energetics after the Fontan operation: contractility-afterload mismatch. J Thorac Cardiovasc Surg. 2003 May;125(5):1061-9. doi: 10.1067/mtc.2003.405. PMID 12771880
- [Background] Tanoue Y, Sese A, Imoto Y, Joh K. Ventricular mechanics in the bidirectional glenn procedure and total cavopulmonary connection. Ann Thorac Surg. 2003 Aug;76(2):562-6. doi: 10.1016/s0003-4975(03)00467-3. PMID 12902104
- [Background] Senzaki H, Masutani S, Ishido H, Taketazu M, Kobayashi T, Sasaki N, Asano H, Katogi T, Kyo S, Yokote Y. Cardiac rest and reserve function in patients with Fontan circulation. J Am Coll Cardiol. 2006 Jun 20;47(12):2528-35. doi: 10.1016/j.jacc.2006.03.022. Epub 2006 May 30. PMID 16781384
- [Background] Cai J, Su Z, Shi Z, Zhou Y, Xu Z, Xu Z, Yang Y. Nitric oxide and milrinone: combined effect on pulmonary circulation after Fontan-type procedure: a prospective, randomized study. Ann Thorac Surg. 2008 Sep;86(3):882-8; discussion 882-8. doi: 10.1016/j.athoracsur.2008.05.014. PMID 18721577